CLINICAL TRIAL: NCT07037199
Title: Efficacy and Safety of Trastuzumab Rezetecan Followed by CDK4/6 Inhibitors and Endocrine Therapy in HR+/HER2-Low/Ultra-Low Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianli Zhao, Breast cancer center, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDE-BRCA
Record Dates: First submitted 2025-06-13; First posted 2025-06-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Advanced Breast Cancer
Keywords: endocrine therapy; breast cancer; Trastuzumab rezetecan; CDK4/6 inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: HR+/HER2-low/ultra-low advanced breast cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR+/HER2-low/ultra-low advanced breast cancer (Experimental): Enrolled patients will be HR+/HER2-low/ultra-low advanced breast cancer patients and receive SHR-A1811 monotherapy for 6-8 cycles until clinical benefit, then transition to dalpiciclib with endocrine therapy until disease progression or unacceptable toxicity.
  Interventions: Drug: Trastuzumab rezetecan + CDK4/6 inhibitors + endocrine therapy

INTERVENTIONS:
Drug: Trastuzumab rezetecan + CDK4/6 inhibitors + endocrine therapy — sequential Trastuzumab rezetecan followed by CDK4/6 inhibitors (Dalpiciclib, Abemaciclib, Ribociclib, Palbociclib) plus endocrine therapy (fulvestrant or aromatase inhibitors)

SUMMARY:
This multicenter, prospective phase II clinical trial evaluates the efficacy and safety of sequential Trastuzumab rezetecan followed by dalpiciclib plus endocrine therapy (fulvestrant or aromatase inhibitors) in 45 patients with HR+/HER2-low/ultra-low advanced breast cancer. Enrolled patients will receive Trastuzumab rezetecan monotherapy for 6-8 cycles until clinical benefit, then transition to CDK4/6 inhibitors with endocrine therapy until disease progression or unacceptable toxicity. The primary endpoint is progression-free survival (PFS), with secondary endpoints including objective response rate (ORR), overall survival (OS), and treatment-related adverse events (TRAEs). The study will be conducted at Sun Yat-sen Memorial Hospital and collaborating centers.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Female patients aged ≥18 years. 2. Pathologically confirmed HER2-low/ultra-low, HR-positive unresectable or metastatic breast cancer:

1. HER2-low: IHC 1+ or IHC 2+/ISH-negative；HER2-ultra-low: IHC 0 with membranous staining (>0 but <1+). HR+: ≥10% tumor cells with ER/PR nuclear staining (verified by central pathology review).
2. Disease stage: Recurrent/metastatic disease; locally recurrent cases must be deemed unresectable by investigators.

3. Prior therapy:

1. Disease progression after endocrine therapy (ET) + CDK4/6 inhibitor in the advanced/metastatic setting.
2. Progression within 12 months of adjuvant ET + CDK4/6 inhibitor allowed.
3. ≤1 line of prior ET and ≤1 line of chemotherapy for advanced disease. 4. Measurable disease per RECIST 1.1 (including lytic/mixed bone-only metastases).

5. ECOG PS 0-1. 6. Adequate organ function (no transfusions/G-CSF within 2 weeks prior):

1. Hematologic: ANC >1.5×10⁹/L; platelets >90×10⁹/L; Hb >90 g/L.
2. Hepatic: Total bilirubin ≤ULN (≤2×ULN if Gilbert's syndrome). ALT/AST ≤1.5×ULN (≤5×ULN with liver metastases). Alkaline phosphatase ≤2.5×ULN.
3. Renal: BUN/Cr ≤1.5×ULN.
4. Cardiac: LVEF ≥50%;
5. QTcF <470 ms. 7. Voluntary participation with signed informed consent.

Exclusion Criteria:

Participants will be excluded if they meet any of the following conditions:

1. Prior anti-HER2 therapy at any stage (including HER2-ADCs such as T-DM1 or T-DXd).
2. Significant cardiac disease, including:

1) Heart failure or systolic dysfunction (LVEF <50%). 2) High-risk/treated angina or arrhythmias (e.g., Type II Mobitz II/third-degree AV block, ventricular tachycardia).

3) Clinically significant valvular disease. 4) ECG-confirmed transmural myocardial infarction. 5) Uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg). 3. Interstitial lung disease (ILD)/pneumonitis:

1. History of non-infectious ILD requiring steroids.
2. Current ILD or suspected ILD that cannot be ruled out by imaging at screening. 4. Impaired drug absorption due to:

1) Dysphagia, chronic diarrhea, intestinal obstruction, or other factors affecting oral medication intake.

5. Uncontrolled third-space effusions (e.g., pleural/peritoneal effusions) not manageable by drainage.

6. Pregnancy, lactation, or unwillingness to use effective contraception during and for 7 months post-treatment.

7. Other exclusions:

1. Severe comorbidities interfering with treatment (e.g., active HBV, pulmonary infections requiring therapy).
2. Any condition deemed unsuitable by investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2-year PFS
  Progression-free survival rate at 2 years, calculated from the date of randomization to the first documented disease progression (per RECIST 1.1) or death due to any cause, whichever occurred first

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | ORR (CR+PR rate per RECIST 1.1) with ≥30% tumor reduction at 2 years post-enrollment, assessed by investigators
  The proportion of patients achieving ≥30% reduction in tumor volume (sum of complete response [CR] and partial response [PR] rates) during the 2-year follow-up period, assessed from enrollment. The primary endpoint is the percentage of patients with ≥30% tumor shrinkage, as evaluated by investigators per RECIST 1.1 criteria
Clinical Benefit Rate (CBR) | CBR (CR+PR+SD≥24 weeks rate per RECIST 1.1) at 2 years post-enrollment, assessed by investigators.
  The proportion of patients achieving either ≥30% tumor reduction or maintaining stable disease (SD) for ≥24 weeks during the 2-year follow-up period (sum of complete response [CR], partial response [PR], and SD lasting ≥24 weeks), as assessed by investigators according to RECIST 1.1 criteria
Disease Control Rate (DCR) | DCR (CR+PR+SD rate per RECIST 1.1) at 2 years post-enrollment (investigator-assessed)
  The proportion of patients achieving tumor stabilization or reduction (sum of complete response [CR], partial response [PR], and stable disease [SD] rates) during the 2-year follow-up period from enrollment, as assessed by investigators per RECIST 1.1 criteria
Overall Survival (OS) | OS (time from enrollment to death) at 2-year follow-up (primary endpoint)
  The time from enrollment to death from any cause during the 2-year follow-up period, with the primary endpoint being the duration from randomization to death event
Treatment-Related Adverse Events (TRAEs) | TRAEs (all AEs from first dose to 30 days post-treatment) graded by CTCAE v5.0, with causality assessment
  All adverse events (AEs) occurring from enrollment until treatment discontinuation during the 2-year follow-up period, including their type, incidence rate, severity grade (assessed per NCI-CTCAE v5.0 criteria), seriousness, and relationship to the study treatment.
Quality of Life (QoL) | QoL (EORTC QLQ-C30) evaluated serially from baseline to treatment discontinuation over 2 years
  Assessed using the EORTC QLQ-C30 questionnaire at baseline (enrollment), during each efficacy evaluation timepoint, and at treatment discontinuation throughout the 2-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: JianLi Zhao, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No